CLINICAL TRIAL: NCT01801267
Title: A Randomized Controlled Trial of Endoscopic Third Ventriculostomy Versus Ventricular Shunt for Children With Communicating Hydrocephalus
Brief Title: Third Ventriculostomy Versus Shunt for Children With Hydrocephalus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pediatric Hydrocephalus Foundation (Unknown); Children's Miracle Network Hospitals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043098
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Communicating Hydrocephalus
Keywords: Hydrocephalus; Pediatric; Ventricular shunt; Ventriculoperitoneal shunt; Third ventriculostomy; Randomized controlled trial
MeSH Terms: conditions — Hydrocephalus | interventions — Ventriculostomy; Cerebrospinal Fluid Shunts; Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic third ventriculostomy (ETV) (Experimental): Pediatric patients in need of CSF-diversion surgery will undergo an endoscopic third ventriculostomy (ETV).
  Interventions: Procedure: Endoscopic third ventriculostomy (ETV)
- Ventricular shunt (Active Comparator): Pediatric patients in need of CSF-diversion surgery will undergo ventricular shunt placement or revision.
  Interventions: Procedure: Ventricular shunt

INTERVENTIONS:
Procedure: Endoscopic third ventriculostomy (ETV) — Pediatric patients in need of CSF-diversion surgery will undergo an endoscopic third ventriculostomy (ETV). A neurosurgeon will make a small hole in the third ventricle (a fluid space in the brain) to allow CSF to flow out of the ventricles.
  Other Names: ETV; third ventriculostomy
  Arms: Endoscopic third ventriculostomy (ETV)
Procedure: Ventricular shunt — Pediatric patients in need of CSF-diversion surgery will undergo ventricular shunt placement or revision. A neurosurgeon will insert a small tube into the ventricle (a fluid space in the brain) and connect this tube to another location in the body so that CSF can flow out of the brain and be absorbed elsewhere in the body - the belly, the top of the heart or the side of the lung. If a patient already has a shunt which is not working, a neurosurgeon will fix or replace it. This will serve as the Control arm of the study.
  Other Names: VP shunt; VA shunt; ventriculoperitoneal shunt; ventriculoatrial shunt; ventriculopleural shunt
  Arms: Ventricular shunt

SUMMARY:
Ventriculoperitoneal shunts are the standard of care for patients with communicating hydrocephalus, but they have a high failure rate - up to 40% fail within 1 year and 50% fail within 2 years. It has long been assumed that endoscopic third ventriculostomy (ETV) would not work in this population and is better suited to patients with obstructive hydrocephalus (such as from a tumor blocking cerebral-spinal fluid (CSF) pathways). However, as scientists learn more about CSF and the way our brains absorb this fluid, they have learned that this may not be so straight-forward. Recent small studies have shown that ETVs can work in a good percentage of children with communicating hydrocephalus, too. But no randomized controlled trials have been done to compare these two treatments directly to determine which will provide children with a better prognosis, fewer surgeries over their lifetime, less time in the hospital and the greatest chance at as normal a life as possible.

The investigators will conduct a trial to compare these two surgical treatments where patients will be randomized to receive either a shunt or an ETV. Because ETV has been shown to have a high failure rate in newborns, the investigators will not include these patients and instead will study patients who come to Duke University with communicating hydrocephalus between the ages of 1 year and 18 years. The study will include patients with ventricular shunts who are in need of revision and patients who were just diagnosed and need their first shunt.

All patients who agree to participate will be randomized to receive either an ETV or a shunt. The study team will follow them for one year from the time of the surgery and will determine what percentage of patients require further CSF-related surgeries, how long they go after their surgery before they need another surgery, how much time they spend in the hospital and what percentage of patients suffer CSF-infections or other problems related to the surgery or their hydrocephalus. The study team will examine these results and determine if ETV is a safer or more effective treatment for children with communicating hydrocephalus than is a ventricular shunt.

ELIGIBILITY:
Inclusion Criteria:

* Children age 1-18 years
* Patients with communicating hydrocephalus who present in need of CSF diversion surgery, as diagnosed by radiographic imaging (CT or MRI of brain) as well as clinical signs or symptoms of increased intracranial pressure
* Informed consent according to institutional guidelines must be obtained from each patient's parent or legal guardian, or by the patient him/herself if he/she is 18 years of age

Exclusion Criteria:

* An active Central Nervous System malignancy (cancer)
* The presence of two or more current ventricular catheters indicating that the ventricles do not communicate with each other
* The inability of the parent/guardian or patient to provide informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time until need for further CSF-related surgeries | one year
  The measurement will be the time between the initial randomized study surgery and any additional CSF-related surgery that the patient needs for a maximum of one year.

SECONDARY OUTCOMES:
Total number of CSF-related surgeries needed within one year | one year
  The measurement will be the total number of CSF-related surgeries that a patient requires within one year of their initial randomized study surgery.

OTHER OUTCOMES:
Morbidities | one year
  The measurement will be the percentage of patients who suffer CSF-infections or other problems related to the surgery or their hydrocephalus within one year after their initial randomized surgery.
Time spent in the hospital | one year
  The measurement will be how much time patients in each group spend in the hospital during the one year after their initial randomized surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie R Muh, MD, MS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No